CLINICAL TRIAL: NCT07207343
Title: To Evaluate the Safety and Efficacy of Ultrasound-guided HIFU for the Symptom Relief of Inoperable Abdominal Tumors.
Brief Title: Symptomatic Abdominal Tumors Are Unsuitable for Surgical Resection, High-intensity Focused Ultrasound (HIFU) Treatment Will be Applied to the Tumors. Postoperatively, Continuous Evaluation and Analysis of the Ablation Effect Will be Performed Using CT or MRI Imaging.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202309073DIPB
Record Dates: First submitted 2025-10-01; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Liver Cancer; HIFU
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- symptomatic abdominal tumors who are unsuitable for surgical resection (Experimental)
  Interventions: Device: Haifu Focused Ultrasound tumor therapeutic System

INTERVENTIONS:
Device: Haifu Focused Ultrasound tumor therapeutic System — Haifu Focused Ultrasound tumor therapeutic System is a tumor ablation technique developed in recent years that allows for non-invasive treatment of solid tumors using High-Intensity Focused Ultrasound (HIFU). This method works by physically focusing ultrasound energy at a single point within biological tissue, creating a focal zone of high-power, low-frequency ultrasound that induces mechanical fragmentation (histotripsy) and cavitation effects, dissolving the tissue into fragments and destroying tumor cells. Under real-time ultrasound imaging guidance, various scanning treatment protocols are used to move the focal point throughout the treatment zone, effectively ablating the tumor tissue. The destroyed tumor tissue is gradually absorbed by the body. Since this technique does not require needle puncture, electrode insertion, radiation, or thermal effects, it is minimally invasive and holds the potential to overcome the limitations of existing ablation technologies.

SUMMARY:
Solid tumors may cause symptoms such as pain due to compression or space-occupying effects. For patients unsuitable for surgical resection, the primary clinical recommendation for malignant tumors is chemotherapy or local radiotherapy to delay tumor progression, improve quality of life, and extend survival. For benign tumors, however, there are currently no effective alternative recommendations. For unresectable tumors, local ablation therapies such as radiofrequency ablation (RFA) are considered potential curative options. Nonetheless, the major limitations of RFA include its invasive puncture procedure, which may lead to bleeding or needle-track tumor seeding, and its reduced efficacy for tumors located adjacent to blood vessels, thereby restricting its use mainly to small hepatocellular carcinomas.

High-Intensity Focused Ultrasound (HIFU) is an emerging ablation tool developed in recent years that provides non-invasive treatment for solid tumors. Its therapeutic principle involves focusing ultrasound waves onto a single point within biological tissue, where the concentrated energy generates thermal, mechanical, and cavitation effects that destroy tumor cells. Under real-time monitoring with ultrasound imaging systems, the focal point can be moved across the treatment area through various scanning approaches, thereby ablating the targeted tumor tissue. The ablated tissue will gradually be absorbed and replaced by fibrosis within the body. Since HIFU does not require needle puncture into the body, it is considered non-invasive.

This clinical trial will employ the Haifu Focused Ultrasound Tumor Therapeutic System, which was approved and registered by the Taiwan Ministry of Health and Welfare in 2012 for the ablation of uterine fibroids. The proposed study targets patients with intra-abdominal benign or malignant tumors who are unsuitable for surgical resection but present with tumor-related symptoms. Tumors will be treated with HIFU, postoperative complications will be monitored, treatment response will be evaluated one month after therapy, and patient survival will be followed up to verify the clinical feasibility and safety of this system.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 20 years.
2. Ability to understand and comply with the routine care requirements of this trial and provide signed informed consent.
3. Patients with intra-abdominal tumors measuring 3-10 cm in diameter, such as hepatobiliary and pancreatic cancers, or benign/malignant retroperitoneal tumors, who present with tumor-related symptoms or discomfort.
4. Patients deemed unsuitable for surgical resection due to distant metastasis, vascular or vital organ invasion, or the high risk of impaired organ function if resection were performed.
5. Good general condition with an ECOG (Eastern Cooperative Oncology Group) performance status of 0-1, and an ASA (American Society of Anesthesiology) score < 3.
6. No severe hepatic or renal dysfunction (Child-Pugh class A/B); total bilirubin ≤ 5 mg/dL; ALT and AST ≤ 5 × upper limit of normal; serum creatinine ≤ 2 × upper limit of normal.
7. Normal coagulation function: PT-INR ≤ 2.0, platelet count ≥ 100,000.
8. Estimated survival of more than 3 months.
9. Maximum tumor depth from skin surface ≤ 11 cm.

Exclusion Criteria:

1. Tumors that cannot be clearly localized under ultrasound examination.
2. No safe acoustic pathway for ultrasound to reach the tumor site upon imaging evaluation, such as when the pathway includes skin scars, bowel gas, calcified tumors, or bones that interfere with ultrasound transmission.
3. Pregnant women.
4. Participation in any other tumor-related clinical trial within 30 days prior to treatment.
5. Radiotherapy to the focused ultrasound treatment area within 30 days before or after treatment.
6. Presence of arterial calcification within the treatment area.
7. Requirement for systemic pharmacological treatment within two weeks before or after the procedure.
8. Deemed unsuitable for treatment by the principal investigator.
9. Presence of surgically related metallic implants in the body.
10. Inability to undergo CT/MRI examinations.
11. Other contraindications related to the investigational device:

    1. Poor tolerance to anesthetic agents
    2. Target tumor located less than 1 cm from the skin surface
    3. Severe dysfunction of vital organs (heart, liver, kidney, brain, or lung)
    4. Severe systemic disorders, extreme fatigue, or significant ascites
    5. Severe diabetes mellitus
    6. Presence of skin ulceration or impending ulceration
    7. Target lesion involving major vessels or portal vein thrombosis, or tumors invading vessel walls or causing significant vascular compression
    8. Tumor invasion into the gastrointestinal or respiratory tract
    9. Tumor with active infection, unless the infection has been controlled
    10. Patients with severe collagenosis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
VAS with preoperative baseline within six months | six months
  The main goals are to confirm if the quality of life of subjects improves after treatment with a focused ultrasound system and to assess the safety of the treatment. VAS score measures pain intensity using a 10-cm line with "no pain" at 0 point and "worst possible pain" at 10 points.
SF-36 with preoperative baseline within six months | six months
  The main goals are to confirm if the quality of life of subjects improves after treatment with a focused ultrasound system and to assess the safety of the treatment. SF-36 score range from 0 to 100, with higher scores indicating better health

SECONDARY OUTCOMES:
Comparison of Tumor Volume Before and After Treatment | six months
  Comparison of tumor volume changes before and after treatment with the focused ultrasound system using CT/MRI imaging, based on RECIST criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan